CLINICAL TRIAL: NCT02745704
Title: The Optimizing Treatment of PegIFN Alfa in HBeAg-negative Chronic Hepatitis B Patients With Low Level HBsAg
Brief Title: The Optimizing Treatment of PegIFN Alfa in HBeAg-negative CHB Patients With Low Level HBsAg
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: Peking University (Other); Huazhong University of Science and Technology (Other); Nanchang University (Other); Huizhou Municipal Central Hospital (Other); First People's Hospital, Shunde China (Other); Shenzhen Third People's Hospital (Other); First People's Hospital of Foshan (Other); Tang-Du Hospital (Other); First Affiliated Hospital of Kunming Medical University (Other); Yuebei People's Hospital (Other)
Responsible Party: Principal Investigator, Zhiliang Gao, chief director of department of infectious disease, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3rd-SYSU-I-Cure
Record Dates: First submitted 2016-04-11; First posted 2016-04-20 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Chronic Hepatitis B
Keywords: chronic hepatitis B; peginterferon alfa
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PEG-IFN group (Experimental): Hepatitis B e antigen (HBeAg)-negative CHB patients who had received NAs for more than 12 months, with HBsAg <1500 IU/ mL and Hepatitis B virus DNA not detectable, are to receive peginterferon alfa-2a 180 micrograms/week or peginterferon alfa-2b 80 micrograms/week for 48 weeks.
  Interventions: Drug: Peginterferon alfa
- NAs group (No Intervention): Patients do not need to change their NAs treatment.

INTERVENTIONS:
Drug: Peginterferon alfa — peginterferon alfa-2b 80 micrograms/week or peginterferon alfa-2a 180 micrograms/week
  Arms: PEG-IFN group

SUMMARY:
As HBsAg clearance is uncommon in chronic hepatitis B (CHB) patients on nucleoside analogues (NAs) therapy. The purpose of this study is to optimize HBsAg clearance in CHB Patients with sequential treatment of pegylated interferon alpha and NAs.

DETAILED DESCRIPTION:
In order to optimize HBsAg clearance in CHB patients with low level HBsAg, the investigators enrolled patients who had received, and responded to, NAs for more than 12 months(see the inclusion criteria), and patients are switched to receive peginterferon alfa-2a 180 micrograms/week or peginterferon alfa-2b 80 micrograms/week for 48 weeks and follow up for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. CHB patients who had received NAs for more than 12 months.
2. Hepatitis B e antigen (HBeAg)-negative and anti-HBeAg positive.
3. Hepatitis B surface antigen (HBsAg) positive and <1500 IU/mL.
4. Hepatitis B virus DNA not detectable(Roche Cobas).

Exclusion Criteria:

1. Patients with liver cirrhosis, Hepatocellular Carcinoma or other malignancies.
2. Patients with other factors causing liver diseases.
3. Pregnant and lactating women.
4. Patients with concomitant HIV infection or congenital immune deficiency diseases.
5. Patients with diabetes, autoimmune diseases.
6. Patients with important organ dysfunctions.
7. Patients with serious complications (e.g., infection, hepatic encephalopathy, hepatorenal syndrome, gastrointestinal bleeding.)
8. Patients who receive antineoplastic or immunomodulatory therapy in the past 12 months.
9. Patients who can't come back to clinic for follow-up on schedule.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-04; Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
HBsAg Clearance | 72 weeks
  Percentage of Participants with HBsAg negative.
HBsAg Seroconversion | 72 weeks
  Percentage of Participants with HBsAg negative and anti-HBsAg positive.

CONTACTS AND LOCATIONS:
Locations (1):
- The third affiliated hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided